CLINICAL TRIAL: NCT07269262
Title: Feasibility and Acceptability of a Mobile Application "SUPPORT-T" to Increase Equitable Access to Palliative Care in Patients With Progressive Pulmonary Fibrosis (PPF) and Their Caregivers
Brief Title: SUPPORT-T in Patients With Progressive Pulmonary Fibrosis and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kathleen Lindell, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00146761
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: Progressive Pulmonary Fibrosis; Interstitial Lung Disease
Keywords: Education; Interstitial Lung Disease (ILD)
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SUPPORT-T Intervention Arm (Experimental): Participants in the intervention arm will have a telehealth preparatory visit scheduled 1 week later (Week 2) with the Study Coordinator and will be provided with the study number to call with questions.
  SUPPORT-T will be delivered biweekly at TeleHealth Visits 1-4 via a secure interface via MUSC telehealth platform. The nurse interventionist will receive results from the REDCap survey after each TH visit and contact the patient biweekly after each TH visit using the MUSC Telehealth and/or Health platform. The nurse interventionist will be available for any questions and communicate with the participants via bi-directional texts (SC will maintain a log of those texts).
  • All participants will complete questionnaires at Week 1, Week 9, Month 6, and Month 12
  Interventions: Other: SUPPORT-T Educational Intervention
- Enhanced Usual Care Control Group (No Intervention): * Participants in the enhanced usual care arm will receive printed education materials from the Pulmonary Fibrosis Foundation (PFF) and the nurse interventionist's contact information.
  * All participants will complete questionnaires at Week 1, Week 9, Month 6, and Month 12

INTERVENTIONS:
Other: SUPPORT-T Educational Intervention — SUPPORT-T will be delivered biweekly at TeleHealth Visits 1-4 via a secure interface via MUSC telehealth platform. The nurse interventionist will receive results from the REDCap survey after each TH visit and contact the patient biweekly after each TH visit using the MUSC Telehealth and/or Health platform. The nurse interventionist will be available for any questions and communicate with the participants via bi-directional texts (SC will maintain a log of those texts)
  Arms: SUPPORT-T Intervention Arm

SUMMARY:
This pilot randomized controlled trial evaluates the feasibility, acceptability, and accessibility of SUPPORT-T, a digitally delivered palliative care intervention for patients with Progressive Pulmonary Fibrosis (PPF) and their caregivers. The intervention includes a 9-week digital application guided by a nurse interventionist and quarterly virtual support groups over one year. Participants will be recruited from rural South Carolina and urban New York City. The study compares SUPPORT-T to Enhanced Usual Care and aims to inform a future multi-site trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Confirmed diagnosis of PPF
* English or Spanish speaking

Caregiver Inclusion Criteria:

* adult, ≥ 18 years old
* Designated and identified by patient as providing most of the emotional, financial, and/or physical support (i.e., the individual most involved in care, does not have to live with patient)
* Able to speak and understand English.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Disease Preparedness | 10 months
  Feasibility outcomes include number of participants recruited weekly, number of participants who declined, and number of participants who did not meet eligibility requirements, data collection procedures, and participant responses. Feasibility data will inform future studies on approaches for recruitment and retention, study procedures, and timing and participant capacity to complete surveys/interviews.
Disease Preparedness Feasibility | 10 months
  Feasibility outcomes include number of participants recruited weekly, number of participants who declined, and number of participants who did not meet eligibility requirements, data collection procedures, and participant responses. Feasibility data will inform future studies on approaches for recruitment and retention, study procedures, and timing and participant capacity to complete surveys/interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes